CLINICAL TRIAL: NCT01166438
Title: Efficacy and Impact of Botulinum Toxin A Versus Anticholinergic Therapy for the Treatment of Bothersome Urge Urinary Incontinence
Brief Title: Anticholinergic vs. Botox Comparison Study
Acronym: ABC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PFDN 17; 2U01HD041249 (NIH); 2U10HD041250 (NIH); 2U10HD041261 (NIH); 2U10HD041267 (NIH); 1U10HD054136 (NIH); 1U10HD054214 (NIH); 1U10HD054215 (NIH); 1U10HD054241 (NIH)
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Urge Urinary Incontinence; Overactive Bladder
Keywords: incontinence; overactive bladder; botox; anticholinergic
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; Solifenacin Succinate; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox A (Experimental): A single intradetrusor injection of 100U botulinum toxin A (Botox A®) plus daily oral placebo tablets
  Interventions: Drug: Botulinum toxin A (Botox A®)
- Standardized Anticholinergic Regimen (Active Comparator): A standardized 3-step anticholinergic regimen of daily oral solifenacin 5mg, solifenacin 10mg, and/or trospium chloride XR 60mg, as well as a single intradetrusor injection of saline (placebo). All subjects will begin on solifenacin 5 mg for 2 mo. If a subject's symptoms are not adequately controlled at 2 mo, she will be escalated to solifenacin 10mg, and similarly at 4 mo to trospium XR 60mg. If a subject's symptoms are adequately controlled on solifenacin 5 mg, she may continue that study medication for the entirety of the study (6 mo). Additionally, if a subject is dose-escalated to solifenacin 10mg at study mo 2 or 4, and her symptoms are adequately controlled, she may continue the solifenacin 10mg dose for the remainder of the study.
  Interventions: Drug: Solifenacin 5mg; Drug: Solifenacin 10mg; Drug: Trospium chloride

INTERVENTIONS:
Drug: Botulinum toxin A (Botox A®) — A single intradetrusor injection of 100U botulinum toxin A in 10 mL plus 0.1 mL of indigo carmine administered during cytoscopy. Between 100 and 200ml of saline is instilled into the bladder prior to injection to allow adequate visualization of the entire bladder urothelium. The treating physician will inject a total of 10.1 mL of the masked substance into approximately 15 to 20 different detrusor muscle sites under direct visualization using disposable needles. Injections will be spread out to equally cover the posterior bladder wall and dome, but spare the bladder trigone and ureteral orifices.
  Other Names: (Botox A®)
  Arms: Botox A
Drug: Solifenacin 5mg — Oral Solifenacin 5mg once a day for up to 6 months
  Other Names: Vesicare
  Arms: Standardized Anticholinergic Regimen
Drug: Solifenacin 10mg — Oral Solifenacin 10mg once a day for up to 4 months
  Other Names: Vesicare
  Arms: Standardized Anticholinergic Regimen
Drug: Trospium chloride — Oral Trospium chloride XR 60mg once a day for up to 2 months
  Other Names: Sanctura
  Arms: Standardized Anticholinergic Regimen

SUMMARY:
Urinary incontinence is a prevalent condition that markedly impacts quality of life and disproportionately affects women. Overactive Bladder syndrome (OAB) is defined as symptoms of urgency and frequency with urge urinary incontinence (OAB-wet) and without urge incontinence (OAB-dry). Conservative first line treatments for urge incontinence combined with other OAB symptoms (OAB-wet) include behavioral therapy, pelvic floor training +/- biofeedback, or the use of anticholinergic medications. These treatment modalities may not result in total continence and often drug therapy is discontinued because of lack of efficacy, side effects and cost or because of not wanting to take a pill. Behavioral therapy and pelvic muscle exercises require consistent, active intervention by the patient which is often not sustained. Thus, the objective of the Anticholinergic vs Botox Comparison Study (ABC) is to determine whether a single intra-detrusor injection of botulinum toxin A (Botox A®) is more effective than a standardized regimen of oral anticholinergics in reducing urge urinary incontinence. The null hypothesis is that there is no difference in the change from baseline in average number of urge urinary incontinence episodes over 6 months between groups.

DETAILED DESCRIPTION:
This study is a 6-month double-blind randomized trial comparing intra-detrusor botulinum toxin A (Botox A®) and anticholinergic therapy in women without neurologic disease with urge incontinence. Subjects will be followed up to an additional six months off study drug to determine duration of treatment effect.

The primary aim is to compare the change in urge incontinence episodes over 6 months between women receiving a single intra-detrusor injection of 100 unit of botulinum toxin A (Botox A®) plus daily oral placebo tablets versus women receiving a single intra-detrusor injection of saline plus daily anticholinergic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed informed consent.
* Females at least 21 years of age
* Five or more urge urinary incontinence episodes on a three-day voiding diary. Urge incontinence episodes will be determined based on voiding diary and subject indication of coincident urge symptoms, allowing self-characterization of incontinence type.
* Urge predominant (urge >50% of total incontinent episodes) urinary incontinence based on self-reported characterization of incontinent episodes on diary.
* Demonstrated ability (or have caregiver demonstrate ability) to perform clean intermittent self-catheterization in the event that this would be required.
* Request for treatment for urge urinary incontinence. The patient may have tried other non-pharmacologic treatments for urge incontinence, such as supervised behavioral therapy, supervised physical therapy, unsupervised physical therapy, supervised biofeedback, and transvaginal electrical stimulation.
* Subject has undergone 3-week washout period if subject were on anticholinergic therapy prior to enrollment.
* Subject is able to complete all study related items and interviews.

Exclusion Criteria:

* Any previous therapy with trospium chloride, solifenacin, or darifenacin
* Failed three or more anticholinergic drugs.
* Contraindication to anticholinergic therapy, specifically with solifenacin or trospium.
* Current symptomatic urinary tract infection that has not resolved prior to randomization.
* Uncontrolled narrow-angle glaucoma
* Gastric retention
* Baseline need for intermittent self catheterization
* PVR >150ml on 2 occasions with void(s) of greater than 150ml
* Surgical treatment for stress incontinence (sling, Burch or urethral injection) or pelvic organ prolapse recommended or planned at enrollment by study investigator(s).
* Any prior intra-detrusor botulinum toxin A injections
* Previous or currently implanted neuromodulation (sacral or tibial).
* Surgically altered detrusor muscle, such as augmentation cystoplasty.
* Known allergy to botulinum toxin A.
* Women with known neurologic disease believed to potentially affect urinary function (Multiple sclerosis, spinal cord injuries, myasthenia gravis, Charcot-Marie-Tooth disease).
* Known allergy to lidocaine.
* Currently pregnant or lactating patients or patients planning pregnancy within the next year.
* Sexually active premenopausal women with a uterus who have either not had a tubal ligation or are not on a medically approved form of contraception for at least 3 months prior to and throughout the duration of the study.
* Cystoscopic findings that preclude injection, in the opinion of the investigator.
* Current or prior bladder malignancy.
* In the opinion of the investigator, inability to understand diary instructions and complete 3-day voiding diary.
* Subjects who are on anticoagulant therapy,excluding aspirin
* Subject has been previously diagnosed with interstitial cystitis or chronic pelvic pain syndrome.
* Subjects with hematuria who have not undergone a clinically appropriate evaluation.
* Subjects taking aminoglycosides at the time of injection.
* Serum creatinine level greater than twice the upper limit of normal within the previous year.
* Two or more hospitalizations for medical conditions in the previous year.
* Plans to move out of area in the next 6 months.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Visco, MD, Study Chair — Duke University
Locations (11):
- United States (11):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - USCD Medical Center, La Jolla, California
  - Kaiser Permanente, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - Oakwood Hospital, Dearborn, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Magee-Women's Hospital, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi BI, Fontes Noronha M, Kaindl J, Wolfe AJ. Complete genome sequences of Aerococcus loyolae ATCC TSD-300T, Aerococcus mictus ATCC TSD-301T, and Aerococcus tenax ATCC TSD-302T. Microbiol Resour Announc. 2024 Jun 11;13(6):e0015624. doi: 10.1128/mra.00156-24. Epub 2024 Apr 23. PMID 38651909
- [Derived] Hendrickson WK, Amundsen CL, Rahn DD, Meyer I, Bradley MS, Smith AL, Myers DL, Jelovsek JE, Lukacz ES. Comparison of 100 U With 200 U of Intradetrusor OnabotulinumToxinA for Nonneurogenic Urgency Incontinence. Female Pelvic Med Reconstr Surg. 2021 Mar 1;27(3):140-146. doi: 10.1097/SPV.0000000000001020. PMID 33620895
- [Derived] Visco AG, Zyczynski H, Brubaker L, Nygaard I, Xu X, Lukacz ES, Paraiso MF, Greer J, Rahn DD, Meikle SF, Honeycutt AA. Cost-Effectiveness Analysis of Anticholinergics Versus Botox for Urgency Urinary Incontinence: Results From the Anticholinergic Versus Botox Comparison Randomized Trial. Female Pelvic Med Reconstr Surg. 2016 Sep-Oct;22(5):311-6. doi: 10.1097/SPV.0000000000000277. PMID 27564385
- [Derived] Visco AG, Brubaker L, Jelovsek JE, Wilson TS, Norton P, Zyczynski HM, Spino C, Sirls L, Nguyen JN, Rahn DD, Meikle SF, Nolen TL; Pelvic Floor Disorders Network. Adherence to Oral Therapy for Urgency Urinary Incontinence: Results from the Anticholinergic Versus Botox Comparison (ABC) Trial. Female Pelvic Med Reconstr Surg. 2016 Jan-Feb;22(1):24-8. doi: 10.1097/SPV.0000000000000215. PMID 26516810
- [Derived] Visco AG, Brubaker L, Richter HE, Nygaard I, Paraiso MF, Menefee SA, Schaffer J, Lowder J, Khandwala S, Sirls L, Spino C, Nolen TL, Wallace D, Meikle SF; Pelvic Floor Disorders Network. Anticholinergic therapy vs. onabotulinumtoxina for urgency urinary incontinence. N Engl J Med. 2012 Nov 8;367(19):1803-13. doi: 10.1056/NEJMoa1208872. Epub 2012 Oct 4. PMID 23036134
- [Derived] Visco AG, Brubaker L, Richter HE, Nygaard I, Paraiso MF, Menefee SA, Schaffer J, Wei J, Chai T, Janz N, Spino C, Meikle S; Pelvic Floor Disorders Network. Anticholinergic versus botulinum toxin A comparison trial for the treatment of bothersome urge urinary incontinence: ABC trial. Contemp Clin Trials. 2012 Jan;33(1):184-96. doi: 10.1016/j.cct.2011.09.019. Epub 2011 Oct 8. PMID 22008247

RESULTS

PARTICIPANT FLOW:
Groups:
- Standardized Anticholinergic Regimen: A standardized 3-step anticholinergic regimen of daily oral solifenacin 5mg, solifenacin 10mg, and/or trospium XR 60mg, as well as a single intradetrusor injection of saline (placebo). All subjects will begin on solifenacin 5 mg for 2 mo. If a subject's symptoms are not adequately controlled at 2 mo, she will be escalated to solifenacin 10mg, and similarly at 4 mo to trospium XR 60mg. If a subject's symptoms are adequately controlled on solifenacin 5 mg, she may continue that study medication for the entirety of the study (6 mo). Additionally, if a subject is dose-escalated to solifenacin 10mg at study mo 2 or 4, and her symptoms are adequately controlled, she may continue the solifenacin 10mg dose for the remainder of the study.
  Solifenacin 5mg: Oral Solifenacin 5mg once a day for up to 6 months
  Solifenacin 10mg: Oral Solifenacin 10mg once a day for up to 4 mon
Period: Double-blind Phase: 1st 6 Months
Arm/Group | Botox A | Standardized Anticholinergic Regimen
Started | 122 | 127
Treated | 121 | 126
Completed | 113 (Completion of 12 month follow-up visit) | 118 (Completion of 12 month follow-up visit)
Not Completed | 9 | 9
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Lost to Follow-up | 0 | 4
Not completed — Not treated | 1 | 1
Period: Off Treatment Follow-up Phase
Arm/Group | Botox A | Standardized Anticholinergic Regimen
Started | 85 | 89
Completed | 51 | 33
Not Completed | 34 | 56
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 4 | 2
Not completed — Lack of Efficacy | 29 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox A | Standardized Anticholinergic Regimen | Total
Number analyzed (Participants) | 121 | 126 | 247
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (10.8) | 56.7 (11.6) | 57.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 126 | 247
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 22 | 44
  Not Hispanic or Latino | 99 | 104 | 203
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 18 | 23 | 41
  White | 96 | 98 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Marital Status [Count of Participants; unit: Participants]
  Married or living as married | 58 | 57 | 115
  Divorced, separated, or widowed | 44 | 48 | 92
  Single, never married | 15 | 16 | 31
  Other | 0 | 1 | 1
  Not reported | 4 | 4 | 8
Educational level at least some college [Count of Participants; unit: Participants] | 86 | 90 | 176
Type of health insurance [Count of Participants; unit: Participants]
  Private only | 61 | 60 | 121
  Medicare or Medicaid only | 10 | 16 | 26
  Other only | 28 | 34 | 62
  Combination of several types | 21 | 16 | 37
  Not reported | 1 | 0 | 1
Smoking status [Count of Participants; unit: Participants]
  Never smoked | 66 | 74 | 140
  Previous smoker | 39 | 40 | 79
  Current smoker | 15 | 12 | 27
  Not reported | 1 | 0 | 1
Menopausal status [Count of Participants; unit: Participants]
  Premenopausal | 15 | 22 | 37
  Postmenopausal | 102 | 92 | 194
  Not sure | 4 | 12 | 16
No prior anticholinergic therapy [Count of Participants; unit: Participants] | 48 | 54 | 102

OUTCOME MEASURES:

1. Primary Outcome: Change in Urge Urinary Incontinence (UUI) Episodes
Description: Change from baseline in mean number of UUI episodes over 6 month double-blind period.
Time Frame: Baseline through 6 months
Measure: Mean (Standard Error); unit: Mean change in UUI episodes from baselin
Arm/Group | Botox A | Standardized Anticholinergic Regimen
Number analyzed (Participants) | 119 | 122
Mean change in UUI episodes from baselin
  1 Month | -3.13 (0.2851) | -3.15 (0.2761)
  2 Months | -3.32 (0.2854) | -3.25 (0.2762)
  3 Months | -3.22 (0.2854) | -3.55 (0.278)
  4 Months | -3.36 (0.2857) | -3.40 (0.2766)
  5 Months | -3.42 (0.2881) | -3.49 (0.2777)
  6 Months | -3.27 (0.2864) | -3.33 (0.2775)

2. Secondary Outcome: Change From Baseline in Score on OABq-SF
Description: Values for the Overactive Bladder Questionnaire Short Form (OABq-SF) are changes from baseline in the adjusted mean scores for months 1 to 6. Scores on the OABq-SF range from 0 to 100, with higher scores on the symptom-severity scale indicating greater severity of symptoms and higher scores on the quality-of-life scale indicating better quality of life. Data were available for 123 participants in the Standardized Anticholinergic Regimen group and 119 in the Botox A A group.
Time Frame: Baseline through 6 months
Measure: Mean (Standard Error); unit: Change from baseline in score on OABq-SF
Arm/Group | Botox A | Standardized Anticholinergic Regimen
Number analyzed (Participants) | 119 | 123
Change from baseline in score on OABq-SF
  OABq-SF Symptom Severity Score | -44.08 (2.54) | -44.55 (2.44)
  OABq-SF Quality of Life Score | 37.13 (2.578) | 37.05 (2.479)

3. Secondary Outcome: Efficacy
Description: Efficacy outcomes assessed reduction and resolution of incontinence, including urgency urinary incontinence (UUI).
Time Frame: 6 months
Population: Efficacy outcomes were assessed in the modified intention-to-treat population, which included all participants who underwent randomization and received a study medication and who had a baseline measure and at least one follow-up measure for the outcome. Proportions were based on data from participants who returned at least four follow-up diaries.
Measure: Count of Participants; unit: Participants
Arm/Group | Botox A | Standardized Anticholinergic Regimen
Number analyzed (Participants) | 112 | 119
Participants
  Complete resolution of UUI | 30 | 16
  Complete resolution of all incontinence | 26 | 13
  >75% reduction in UUI episodes | 61 | 48

4. Secondary Outcome: Change in PFDI-SF and PFIQ-SF Total Scores
Description: Values for Pelvic Floor Distress Inventory Short Form (PFDI-SF) are changes from baseline in the adjusted mean scores for months 3 to 6. Scores on the PFDI-SF range from 0 to 300, with higher scores indicating more symptoms and more bothersome symptoms. Values for the Pelvic Floor Impact Questionnaire Short Form (PFIQ-SF) are changes from baseline in the adjusted mean scores for months 3 to 6. Scores on the PFIQ-SF range from 0 to 300, with higher scores indicating a more negative effect on activities, relationships, and feelings.
Time Frame: Baseline through 6 months
Population: Data were available for 111 participants in the Standardized Anticholinergic Regimen group and 102 in the Botox A group.
Measure: Mean (Standard Error); unit: Changes in adjusted mean scores
Arm/Group | Botox A | Standardized Anticholinergic Regimen
Number analyzed (Participants) | 102 | 111
Changes in adjusted mean scores
  Change from baseline in PFDI-SF total score | -48.20 (5.56) | -43.69 (5.34)
  Change from baseline in PFIQ-SF total score | -33.85 (6.313) | -32.82 (6.065)

5. Secondary Outcome: Patient Global Impression of Improvement
Description: The Patient Global Impression of Improvement (PGI-I) is a patient-reported measure of perceived improvement with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse). Included here are participants who had adequate improvement, defined as a rating of 1 or 2 (much better).
Time Frame: 3 and 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Standardized Anticholinergic Regimen: A standardized 3-step anticholinergic regimen of daily oral solifenacin 5mg, solifenacin 10mg, and/or trospium XR 60mg, as well as a single intradetrusor injection of saline (placebo). All subjects will begin on solifenacin 5 mg for 2 mo. If a subject's symptoms are not adequately controlled at 2 mo, she will be escalated to solifenacin 10mg, and similarly at 4 mo to trospium XR 60mg. If a subject's symptoms are adequately controlled on solifenacin 5 mg, she may continue that study medication for the entirety of the study (6 mo). Additionally, if a subject is dose-escalated to solifenacin 10mg at study mo 2 or 4, and her symptoms are adequately controlled, she may continue the solifenacin 10mg dose for the remainder of the study.
  Solifenacin 5mg: Oral Solifenacin 5mg once a day for up to 6 months
  Solifenacin 10mg: Oral Solifenacin 10mg once a day for up to 4 months
  Trospium chloride: Oral Trospium XR 60mg once a day for up to 2 months
Arm/Group | Botox A | Standardized Anticholinergic Regimen
Number analyzed (Participants) | 111 | 116
Participants
  Month 3 | 61 | 59
  Month 6 | 60 | 67

ADVERSE EVENTS:
Groups:
- Standardized Anticholinergic Regimen: A standardized 3-step anticholinergic regimen of daily oral solifenacin 5mg, solifenacin 10mg, and/or trospium XR 60mg, as well as a single intradetrusor injection of saline (placebo). All subjects will begin on solifenacin 5 mg for 2 mo. Dose escalation or drug change will be based exclusively on the result of the Patient Global Symptom Control Rating. If a subject's symptoms are not adequately controlled at 2 mo, she will be escalated to solifenacin 10mg, and similarly at 4 mo to trospium XR 60mg. If a subject's symptoms are adequately controlled on solifenacin 5 mg, she may continue that study medication for the entirety of the study (6 mo). Additionally, if a subject is dose-escalated to solifenacin 10mg at study mo 2 or 4, and her symptoms are adequately controlled, she may continue the solifenacin 10mg dose for the remainder of the study.
Arm/Group | Botox A | Standardized Anticholinergic Regimen
Serious Adverse Events (participants affected / at risk) | 5/121 | 7/126
Other Adverse Events (participants affected / at risk) | 96/121 | 97/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botox A (N=121) | Standardized Anticholinergic Regimen (N=126)
Cardiac septal hypertrophy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botox A (N=121) | Standardized Anticholinergic Regimen (N=126)
Constipation (Gastrointestinal disorders) | 31 | 37
Diarrhea (Gastrointestinal disorders) | 21 | 15
Dry mouth (Gastrointestinal disorders) | 44 | 64
Nausea (Gastrointestinal disorders) | 6 | 5
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 63 | 74
Chills (General disorders) | 12 | 12
Influenza-like illness (General disorders) | 9 | 7
Injection site pain (General disorders) | 34 | 36
Pyrexia (General disorders) | 8 | 6
Any General Disorders and Administration Site Conditions (General disorders) | 49 | 41
Haematuria (Renal and urinary disorders) | 28 | 23
Urine abnormality (Renal and urinary disorders) | 17 | 14
Urine odour abnormal (Renal and urinary disorders) | 16 | 10
Any Renal and Urinary Disorders (Renal and urinary disorders) | 49 | 38
Dry eye (Eye disorders) | 32 | 31
Any Eye Disorders (Eye disorders) | 34 | 31
Urinary tract infection (Infections and infestations) | 37 | 19
Any Infections and Infestations (Infections and infestations) | 37 | 20
Flank Pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Any Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 11 | 5
Rash (Skin and subcutaneous tissue disorders) | 8 | 6
Any Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 8 | 6
Hypersensitivity (Immune system disorders) | 7 | 1
Any Immune System Disorders (Immune system disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No